CLINICAL TRIAL: NCT04484428
Title: A Phase II, Randomized, Double-blind, Active Comparator, Parallel Group Study to Evaluate the Efficacy and Safety of K-285 Compared With Menthol Gel for the Treatment of Delayed Onset Muscle Soreness (DOMS) in the Lower Extremity
Brief Title: A Study to Evaluate the Efficacy and Safety of K-285 Compared With Menthol Gel for the Treatment of Delayed Onset Muscle Soreness (DOMS) in the Lower Extremity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Internal business decision
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-285-201
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Menthol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A (Experimental): K-285
  Interventions: Drug: K-285
- Treatment Arm B (Active Comparator): Menthol
  Interventions: Drug: Menthol

INTERVENTIONS:
Drug: K-285 — 88 subjects are to be assigned to 1 week dosing, four times a day (QID) (Period 1), and 32 are to be assigned to 3 weeks dosing (Period 1 and Period 2) with 16 subjects each in the two times a day (BID) and QID dosing regimens.
  Arms: Treatment Arm A
Drug: Menthol — 88 subjects are to be assigned to 1 week dosing, four times a day (QID) (Period 1), and 32 are to be assigned to 3 weeks dosing (Period 1 and Period 2) with 16 subjects each in the two times a day (BID) and QID dosing regimens.
  Arms: Treatment Arm B

SUMMARY:
The purpose of this study to evaluate the efficacy and safety of K-285 compared with menthol gel for the treatment of delayed onset muscle soreness (DOMS) in the lower extremity.

ELIGIBILITY:
Inclusion Criteria:

* Subject must provide informed consent before any study-specific evaluation is performed.
* Subject is male and female aged 18 to 35 years, inclusive.
* Subject has a body mass index of 18 to 32 kg/m2, inclusive.
* Subject meets all inclusion criteria outlined in the Clinical Study Protocol.

Exclusion Criteria:

* Subject has a job (e.g., movers, construction workers) that requires regular lifting or involvement of the lower extremities.
* Subject has restless leg syndrome, a chronic pain condition, a history of intermittent claudication, or has taken any medication (e.g., analgesic medication, sleep medication, muscle relaxant, anticonvulsant, or antidepressant) in the last 6 months to treat a chronic pain condition, or has another painful physical condition in a lower extremity that, in the opinion of the investigator, may confound study assessments.
* Subject has received oral or topical analgesic medications within 14 days before the Screening Visit.
* Subject meet any other exclusion criteria outlined in the Clinical Study Protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Research, LLC, Pasadena, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants underwent pre- and post-exercise evaluations, as well as other screening assessments, to determine eligibility for randomization. Those qualifying were randomly assigned in a 1:1 ratio to Treatment Arm A (K-285 gel) or Treatment Arm B (Menthol gel). All baseline, endpoint, and safety analyses were conducted based on the treatment arm participants were randomized to. Participants not qualifying for randomization were given appropriate standard of care.
Groups:
- K-285: K-285 gel for up to 3 weeks based on pre-specified treatment assignments.
- Menthol: Menthol gel for up to 3 weeks based on pre-specified treatment assignments.
Period: Overall Study
Arm/Group | K-285 | Menthol
Started | 63 | 63
Completed | 56 | 60
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: * Participants were randomly assigned to Treatment Group A (K-285 gel) or Treatment Group B (Menthol gel). Analyses were conducted based on the treatment group participants were randomized to.
  * Demographics and baseline characteristics including identification of the study leg and baseline pain intensity were presented by-subject and summarized overall and by treatment group using FAS.
  * All 126 participants (100.0%) were included in the FAS, PPS, and Safety Set populations.
Units Other Than Participants: Legs
Groups:
- Total: Total of all reporting groups
Arm/Group | K-285 | Menthol | Total
Number analyzed (Participants) | 63 | 63 | 126
Number analyzed (Legs) | 126 | 126 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (4.89) | 27.2 (4.39) | 27.8 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 61
  Male | 33 | 32 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 45
  Not Hispanic or Latino | 41 | 40 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 14 | 11 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 18 | 28
  White | 39 | 30 | 69
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Qualifying (Baseline) eVAS Score for Study Leg while Standing [Mean (Standard Deviation); unit: Points] — Visual Analog Scale (VAS), a unidimensional measure of pain intensity, is a continuous scale from 0 to 100 comprised of a horizontal line anchored by 2 descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst possible pain" (score of 100). The pain eVAS was electronically displayed and was completed by the study participant. The integers of the eVAS were referred to as points. Population: The analysis was based on participants' self-reported pain intensity scores in the study leg.
  Points
    number analyzed (Legs) | 63 | 63 | 126
    (all) | 71.4 (13.94) | 69.1 (13.58) | 70.2 (13.76)
Qualifying (Baseline) eVAS Score for Study Leg at Rest [Mean (Standard Deviation); unit: Points] — Visual Analog Scale (VAS), a unidimensional measure of pain intensity, is a continuous scale from 0 to 100 comprised of a horizontal line anchored by 2 descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst possible pain" (score of 100). The pain eVAS was electronically displayed and was completed by the study participant. The integers of the eVAS were referred to as points. Population: The analysis was based on participants' self-reported pain intensity scores in the study leg.
  Points
    number analyzed (Legs) | 63 | 63 | 126
    (all) | 62 (15.14) | 57.5 (15.51) | 59.8 (15.43)
Qualifying (Baseline) eVAS Score for Non-Study Leg while Standing [Mean (Standard Deviation); unit: Points] — Visual Analog Scale (VAS), a unidimensional measure of pain intensity, is a continuous scale from 0 to 100 comprised of a horizontal line anchored by 2 descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst possible pain" (score of 100). The pain eVAS was electronically displayed and was completed by the study participant. The integers of the eVAS were referred to as points. Population: The analysis was based on participants' self-reported pain intensity scores in the non-study leg.
  Points
    number analyzed (Legs) | 63 | 63 | 126
    (all) | 69.8 (16.77) | 68.2 (16.38) | 69 (16.53)
Qualifying (Baseline) eVAS Score for Non-Study Leg at Rest [Mean (Standard Deviation); unit: Points] — Visual Analog Scale (VAS), a unidimensional measure of pain intensity, is a continuous scale from 0 to 100 comprised of a horizontal line anchored by 2 descriptors, one for each symptom extreme: "no pain" (score of 0) and "worst possible pain" (score of 100). The pain eVAS was electronically displayed and was completed by the study participant. The integers of the eVAS were referred to as points. Population: The analysis was based on participants' self-reported pain intensity scores in the non-study leg.
  Points
    number analyzed (Legs) | 63 | 63 | 126
    (all) | 59.1 (18.77) | 54.7 (19.44) | 56.9 (19.16)

OUTCOME MEASURES:

1. Primary Outcome: Sum of Pain Intensity Difference Between 0 to 24 Hours (SPID0-24) for Study Leg While Standing
Description: * Pain Intensity (PI) was assessed for study leg while standing using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 24 hours after initiating treatment (SPID24). SPID24 derived from pain scores assessed over 24 hours on a 0 -100 point scale. SPID24 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 24 Hours
Population: * Subjects in each treatment Arm/Group (K-285 and Menthol Gel) received intervention based on pre-specified treatment assignments
  * Baseline and Endpoint analysis were performed and presented by treatment Arms/Groups.
  * Demographics and baseline characteristics are presented in a by-subject listing and summarized overall and by treatment Arm using the FAS.
  * All 126 participants (100.0%) were included in the FAS, the PPS, and Safety populations.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Groups:
- Menthol Gel: Menthol gel for up to 3 weeks based on pre-specified treatment assignments
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -488.0 (58.54) | -512.0 (58.53)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.773, ANCOVA

2. Secondary Outcome: SPID0-24 at Rest for Study Leg
Description: * Pain Intensity (PI) was assessed at rest for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 24 hours after initiating treatment (SPID24). SPID24 derived from pain scores assessed over 24 hours on a 0 -100 point scale. SPID24 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 24 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -358.3 (54.42) | -355.6 (54.45)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.972, ANCOVA

3. Secondary Outcome: SPID0-12 While Standing for Study Leg
Description: * Pain Intensity (PI) was assessed while standing for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 12 hours after initiating treatment (SPID12). SPID12 derived from pain scores assessed over 12 hours on a 0 -100 point scale. SPID12 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 12 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -190.2 (26.83) | -209.2 (26.83)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.617, ANCOVA

4. Secondary Outcome: SPID0-12 at Rest for Study Leg
Description: * Pain Intensity (PI) was assessed at rest for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 12 hours after initiating treatment (SPID12). SPID12 derived from pain scores assessed over 12 hours on a 0 -100 point scale. SPID12 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 12 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -131.5 (25.28) | -140.8 (25.29)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.796, ANCOVA

5. Secondary Outcome: SPID0-48 While Standing for Study Leg
Description: * Pain Intensity (PI) was assessed while standing for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 48 hours after initiating treatment (SPID48). SPID48 derived from pain scores assessed over 48 hours on a 0 -100 point scale. SPID48 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 48 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -1229.9 (123.15) | -1221.1 (123.14)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.960, ANCOVA

6. Secondary Outcome: SPID0-48 at Rest for Study Leg
Description: * Pain Intensity (PI) was assessed at rest for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 48 hours after initiating treatment (SPID48). SPID48 derived from pain scores assessed over 48 hours on a 0 -100 point scale. SPID48 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 48 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -959.4 (114.80) | -909.5 (114.85)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.761, ANCOVA

7. Secondary Outcome: SPID0-72 While Standing for Study Leg
Description: * Pain Intensity (PI) was assessed while standing for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 72 hours after initiating treatment (SPID72). SPID72 derived from pain scores assessed over 72 hours on a 0 -100 point scale. SPID72 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 72 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -2154.1 (184.65) | -2160.8 (184.64)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.979, ANCOVA

8. Secondary Outcome: SPID0-72 at Rest for Study Leg
Description: * Pain Intensity (PI) was assessed at rest for study leg using a patient rated 0-100 point scale where 0 = 'no Pain' and 100 = 'worst possible pain. Pain Intensity Differences (PID) was the difference between PI at time (i) minus PI at time (t+1). The Sum of Pain Intensity Difference (SPID) was calculated as a time-weighted Sum of PID scores over a number of hours.
  * Sum of pain intensity differences over 72 hours after initiating treatment (SPID72). SPID72 derived from pain scores assessed over 72 hours on a 0 -100 point scale. SPID72 was computed using the trapezoidal rule, i.e. Σ [T(i+1) - T(i)] x [((PID)(i+1) + PID(i))/2] in an obvious notation, where T(i) is nominal time and PID(i), the pain intensity difference at Time (i).
  * Negative differences correspond to an improvement of pain, while positive differences correspond to recrudescence of pain. A higher negative value of SPID indicates greater pain relief.
Time Frame: Baseline to 72 Hours
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Legs
Arm/Group | K-285 | Menthol Gel
Number analyzed (Participants) | 63 | 63
Number analyzed (Legs) | 63 | 63
score on a scale | -1730.1 (169.61) | -1678.3 (169.68)
Statistical Analysis 1: Comparison: K-285 vs Menthol Gel; Test type: Superiority; p = 0.803, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to 29 Days
Description: * The Safety Set included all participants who had at least 1 study gel application.
  * The safety analyses were conducted based on the treatment group (K-285 or Menthol gel) participants were randomized to.
  * Adverse Event information was assessed according to the treatment Arm/Group and not treatment schedules, as pre-specified in the SAP
  * Treatment emergent adverse events (TEAE) were any adverse event that occurred or worsened after the first dose of study treatment.
Arm/Group | K-285 | Menthol Gel
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 6/63 | 1/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-285 (N=63) | Menthol Gel (N=63)
Application site erythema (General disorders) | 4 | 1
Application site pruritus (General disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Clinical Study Protocol Ver 1.0 (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04484428/Prot_000.pdf
  • Study Protocol: Clinical Study Protocol Ver 2.0 (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT04484428/Prot_001.pdf
  • Statistical Analysis Plan: SAP Interim Analysis (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT04484428/SAP_002.pdf
  • Statistical Analysis Plan: SAP Final (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT04484428/SAP_003.pdf